CLINICAL TRIAL: NCT07366164
Title: The Assisted Fluid Management For High-Risk Patients During Colorectal Surgery: A Randomised Controlled Clinical Trial
Brief Title: Hemodynamic Optimization Using an Artificial Intelligenze System
Acronym: SIMPLY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, RUSSO ANDREA, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 7755
Record Dates: First submitted 2025-09-10; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Hemodynamic (MAP) Stability; Fluid Management

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): fluid therpay fo this grioup will be giuded through the assisted fluid management system
  Interventions: Device: assisted fluid therapy
- control group (No Intervention): patients belonging to this group will receive fluids following a standard hemodynamic protocol

INTERVENTIONS:
Device: assisted fluid therapy — for this intervention, fluids will be administered using an assisted fluid device
  Arms: treatment group

SUMMARY:
This study will investigate the impact of using an automated fluid management system on intraoperative fluid therapy in patients undergoing colorectal surgery. The aim is to evaluate whether automated guidance can optimize hemodynamic stability and reduce the incidence of arterial hypotension,

ELIGIBILITY:
Inclusion Criteria:

- patients >18 years old and ASA 3 scheduled for laparoscopic colorectal surgery

Exclusion Criteria:

* Refusal of consent
* Body Mass Index > 35 kg/m2
* urgent cases
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
amounts of fluids | at the end of surgery
  we registered and compared the amounts of administered fluids after surgery

CONTACTS AND LOCATIONS:
Overall Officials: andrea russo, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Policlinico Gemelli, Roma, RM, Italy